CLINICAL TRIAL: NCT01366404
Title: A Multicenter, Prospective Cohort to Evaluate the Natural History of FFR Guided Percutaneous Coronary Intervention
Brief Title: Study of the Natural History of FFR Guided Percutaneous Coronary Intervention
Acronym: IRIS FFR
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Abbott Medical Devices (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: CVRF2010-09
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
Keywords: FFR
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FFR: Patients who had FFR measurement

SUMMARY:
About 20,000 patients with FFR (Fractional Flow Reserve) will be enrolled and evaluated for the natural history of coronary lesions at 2 years clinical and imaging follow-up.

DETAILED DESCRIPTION:
This is a multicenter, prospective cohort. About 20,000 patients with FFR will be enrolled at multi centres in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 years and older
* FFR measurement on one and more coronary artery stenosis
* Willing and able to provide informed, written consent

Exclusion Criteria:

* Stenosis with TIMI<3 flow
* Graft vessel
* Ejection fraction < 30%
* Angiographic evidence of extreme tortuosity or calcified coronary vessels
* Suspected coronary spasm even after sufficient nitrate injected
* Life expectancy <2 year
* Planned cardiac surgery or planned major non cardiac surgery
* Woman who are breastfeeding, pregnant or planning to become pregnant during the course of the study

Imaging study specific exclusion criteria

* visually-estimated angiographic reference segment diameter of <2.75mm or >4.0mm
* Inappropriate for IVUS/VH/OCT procedures : inability for imaging wire or catheter to pass through the tight stenosis, severe calcification, angulation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had FFR measurement
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2011-06 (Actual); Primary Completion 2037-04 (Estimated); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure | 2 year after index FFR measurement
composite Cardiac Death,Non Fatal Myocardial Infarction, Target Vessel Revascularization, and Indeterminate events | at 2 year after index FFR measurement

SECONDARY OUTCOMES:
Death (all cause and cardiac) | at 2 year after index FFR measurement
MI | at 2 year after index FFR measurement
Target vessel revascularization | at 2 year after index FFR measurement
Target lesion revascularization | at 2 year after index FFR measurement
Any re-hospitalization with a cardiac cause | 2 year follow-up after index FFR measurement
cardiac death and myocardial infarction | 2 year follow-up after index FFR measurement
stented lesion related event including death, myocardial infarction, repeat revascularization | 2 year follow-up after index FFR measurement
stroke | 2 year follow-up after index FFR measurement
stent thrombosis | 2 year follow-up after index FFR measurement
anginal status | 2 year follow-up after index FFR measurement
number of anti-anginal medication prescribed | 2 year follow-up after index FFR measurement
complication of FFR measurement | 2 year follow-up after index FFR measurement
clinical predictors of events | 2 year follow-up after index FFR measurement
change in plaque composition (%necrotic core volume) in target segment | 2 year follow-up after index FFR measurement
change in plaque type assessed by VH(Virtual Histology) and OCT(Optical coherence tomography) | 2 year follow-up after index FFR measurement
change in total atheroma volume and percent atheroma volume | 2 year follow-up after index FFR measurement
change in IVUS-measured MLA | 2 year follow-up after index FFR measurement
change in FFR | 2 year follow-up after index FFR measurement

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD,PhD, Principal Investigator — Asan Medical Center
Locations (29):
- South Korea (29):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Chungbuk National University Hospital, Cheongju-si
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National university hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Deajeon St.Mary's hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Ilsan
  - Dong-A Medical Center, Pusan
  - Pusan National University Hospital, Pusan
  - Seoul university Bundang hospital, Seongnam
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung-Hee University Hospital at Kangdong, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahn JM, Park DW, Kim SO, Kang DY, Lee CH, Lee PH, Lee SW, Park SW, Park SJ. Prognostic Value of Resting Distal-to-Aortic Coronary Pressure in Clinical Practice. Circ Cardiovasc Interv. 2020 May;13(5):e007868. doi: 10.1161/CIRCINTERVENTIONS.118.007868. Epub 2020 Apr 29. PMID 32345039
- [Derived] Kang DY, Ahn JM, Kim YW, Moon JY, Lee JS, Koo BK, Lee PH, Park DW, Kang SJ, Lee SW, Kim YH, Park SW, Park SJ. Impact of Coronary Lesion Geometry on Fractional Flow Reserve: Data From Interventional Cardiology Research In-Cooperation Society-Fractional Flow Reserve and Intravascular Ultrasound Registry. Circ Cardiovasc Imaging. 2018 Jun;11(6):e007087. doi: 10.1161/CIRCIMAGING.117.007087. PMID 29895713
- [Derived] Kang DY, Ahn JM, Lee CH, Lee PH, Park DW, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park SJ. Deferred vs. performed revascularization for coronary stenosis with grey-zone fractional flow reserve values: data from the IRIS-FFR registry. Eur Heart J. 2018 May 7;39(18):1610-1619. doi: 10.1093/eurheartj/ehy079. PMID 29529177
- [Derived] Lee JM, Hwang D, Park J, Zhang J, Tong Y, Kim CH, Bang JI, Suh M, Paeng JC, Cheon GJ, Koo BK. Exploring Coronary Circulatory Response to Stenosis and Its Association With Invasive Physiologic Indexes Using Absolute Myocardial Blood Flow and Coronary Pressure. Circulation. 2017 Nov 7;136(19):1798-1808. doi: 10.1161/CIRCULATIONAHA.117.029911. Epub 2017 Aug 29. PMID 28851731
- [Derived] Ahn JM, Park DW, Shin ES, Koo BK, Nam CW, Doh JH, Kim JH, Chae IH, Yoon JH, Her SH, Seung KB, Chung WY, Yoo SY, Lee JB, Choi SW, Park K, Hong TJ, Lee SY, Han M, Lee PH, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park SJ; IRIS-FFR Investigatorsdagger. Fractional Flow Reserve and Cardiac Events in Coronary Artery Disease: Data From a Prospective IRIS-FFR Registry (Interventional Cardiology Research Incooperation Society Fractional Flow Reserve). Circulation. 2017 Jun 6;135(23):2241-2251. doi: 10.1161/CIRCULATIONAHA.116.024433. Epub 2017 Mar 29. PMID 28356440
- [Derived] Lee JM, Kim CH, Koo BK, Hwang D, Park J, Zhang J, Tong Y, Jeon KH, Bang JI, Suh M, Paeng JC, Cheon GJ, Na SH, Ahn JM, Park SJ, Kim HS. Integrated Myocardial Perfusion Imaging Diagnostics Improve Detection of Functionally Significant Coronary Artery Stenosis by 13N-ammonia Positron Emission Tomography. Circ Cardiovasc Imaging. 2016 Sep;9(9):e004768. doi: 10.1161/CIRCIMAGING.116.004768. PMID 27609817
- [Derived] Kang SJ, Ahn JM, Han S, Lee JY, Kim WJ, Park DW, Lee SW, Kim YH, Lee CW, Park SW, Mintz GS, Park SJ. Sex differences in the visual-functional mismatch between coronary angiography or intravascular ultrasound versus fractional flow reserve. JACC Cardiovasc Interv. 2013 Jun;6(6):562-8. doi: 10.1016/j.jcin.2013.02.016. PMID 23787231
- [Derived] Park SJ, Kang SJ, Ahn JM, Shim EB, Kim YT, Yun SC, Song H, Lee JY, Kim WJ, Park DW, Lee SW, Kim YH, Lee CW, Mintz GS, Park SW. Visual-functional mismatch between coronary angiography and fractional flow reserve. JACC Cardiovasc Interv. 2012 Oct;5(10):1029-36. doi: 10.1016/j.jcin.2012.07.007. PMID 23078732